CLINICAL TRIAL: NCT04123782
Title: Focused Shockwave Treatment in the Recovery Process of Acute Muscle Injuries in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Garcia Cugat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REHAB-2019-01
Record Dates: First submitted 2019-07-25; First posted 2019-10-11 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Muscle Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (F-ESWT group) (Active Comparator): 3 sessions, one per week, of electromagnetic focused extracorporeal shockwave treatment (3000 impulses at 0.12 mJ/mm2 per session)
  Interventions: Device: F-ESW Treatment
- Group B (placebo group) (Placebo Comparator): 3 sessions, one per week, of electromagnetic focused extracorporeal shockwave treatment (3000 impulses at 0.01 mJ/mm2 per session)
  Interventions: Device: Placebo F-ESW Treatment

INTERVENTIONS:
Device: F-ESW Treatment — The biological principles on which is based Focused Shockwave Treatment (F-ESWT) is has been demonstrated mostly in terms of improvement of Platelet Derived Growth Factor (PDGF), Vascular Endothelial Growth Factor (VEGF), Fibroblast Growth Factor (FGF), Insulin Growth Factor-1 (IGF-1) and Transforming Growth Factor b1 (TGF-b1).
  Arms: Group A (F-ESWT group)
Device: Placebo F-ESW Treatment — Very low concentration of F-ESW.
  Arms: Group B (placebo group)

SUMMARY:
The biological principles on which is based Focused Shockwave Treatment (F-ESWT) is has been demonstrated mostly in terms of improvement of Platelet Derived Growth Factor (PDGF), Vascular Endothelial Growth Factor (VEGF), Fibroblast Growth Factor (FGF), Insulin Growth Factor-1 (IGF-1) and Transforming Growth Factor b1 (TGF-b1). Nevertheless, to date Focused Shockwave Treatment is not used in the treatment of acute pathologies and consequently in acute muscle lesion, despite there are no contra-indication in that sense. A recent study of Zissler et al. demonstrate how focused shockwave treatment induce an acceleration of the biological process of recovery during the acute phase of muscle injury in rats, and in 2016 Kisch et al. demonstrate that Focused ESWT enhances blood flow in the muscle of rats and repetitive ESWT extended this beneficial effect. The only clinical trial in humans about acute pathology in muscle was realized by Fleckenstein et al. in 2016, in which demonstrate that a single treatment with F-ESWT causes clinically relevant effects in the relief of pain, increase in force and improvement of pain-associated impairments of daily living in subjects affected by DOMS. However, there are no studies in humans that describe the effect of F-ESWT in muscle injuries. Considering the greater number of evidences about the biological effects of F-ESWT, namely anti-inflammation, neo-vascularization and tissue regeneration and their parallelism in many aspects with one of the most novelty treatment of muscle injuries, as for example the growth factors therapy, the hypothesis is to obtain favorable and better outcomes, both ultrasonographic and clinical, in subjects treated with F-ESWT than in subjects treated with standard treatments.

Study Hypothesis: The hypothesis of our study is that 3 sessions of focused shockwave treatment (1 per week), performed in acute phase of injury (≤ 2 weeks), a total of 3.000 shocks with an energy flux density of 0,12 mJ/mm2 at 5 Hz, can improve the recovery process of acute indirect hamstrings injuries, with results both clinical and ultrasonographic.

Primary Objective To analyze the effect of Focused Shockwave Treatment in acute indirect hamstring injuries in soccer players.

Secondary Objectives

* To analyze the effect of Focused Shockwave Treatment in acute indirect hamstring injuries in soccer players.
* To analyze prognostic factors (demographic, clinical, imaging variables).

DETAILED DESCRIPTION:
Primary Objective To analyze the effect of Focused Shockwave Treatment in acute indirect hamstring injuries in soccer players.

Secondary Objectives

* To analyze the effect of Focused Shockwave Treatment in acute indirect hamstring injuries in soccer players.
* To analyze prognostic factors (demographic, clinical, imaging variables). Study Outcome Measures Primary outcome: Repair process, injury size and Return to play Secondary outcomes: Functional scales: VAS, LEFS and Tegner Satisfaction scales: Roles and Maudsley and Likert scale

DESIGN This is a single blind randomized clinical trial that will be conducted in Quirónsalud Barcelona, Spain. The study will enroll patients suffering an acute indirect injury of common tendon of hamstrings, over a 5-months period. The duration of the trial will be of approximately 8 months. This protocol calls for 9 visits to be performed over a 8-weeks period for each patient (see flow-chart). As an intention-to-treat study, data analysis will be based on the randomization of the patients. At Visit 1 (screening visit; T0), patients will first need to provide written signed informed consent before any data is collected or procedures are performed. Then, patients will be screened for eligibility for the study by ascertaining that all inclusion criteria and no exclusion criteria are met. At V1, the Investigator will gather demographic and medical history data and will carry out clinical and ultrasonographic evaluation. The treatment period will consist of three sessions of ESWT, performed one week apart and within 2 weeks from the day of injury. Clinical and ultrasonographic data will continue to be collected during a follow-up period consisting of 9 visits, one per week and performed starting at 1 week from visit 1 (V1;T0). The last follow-up visit will performed at 10 weeks from visit 1 (V1;T0).

Treatment Assignment Procedures i. Randomization Procedures: We will use block randomization, which is commonly used in the two treatment situations where the samples of the two treatments must be equal or equally equal. The process will involve recruiting participants in short blocks and ensuring that half of the participants within each block are assigned to "A" and the other half to "B". Within each block, however, the order of patients will be random. They will be considered blocks of four dimensions: 1. AABB, 2. ABAB, 3. ABBA, 4. BAAB, 5. BABA, 6. BBAA. We will randomly select between these six different blocks for each group of four recruited participants. The random selection will be done using a list of random numbers generated using statistical software (Excel).

ii. Masking Procedures: The participants will be blinded to the type of ESWT treatment and the assessor, data managers, statistician and study monitors will be blinded to the allocation. All participants who receive ESWT treatment will be treated using the same device (Duolith® SD-1 STORZ Medical, Switzerland) regardless of what group they are included in. The participants will not be able to predict the allocated group based on the appearance of the ESWT treatment. The blinding will be maintained until the data are locked. For blinding evaluation, allocation guessing will be assessed immediately after the final treatment. Practitioners and assessors will be instructed to treat the participants according to predefined standard operating procedures during the trial to maintain blinding.

MATERIAL AND METHOD Study intervention

Soccer players suffering from indirect acute hamstring injury, will be selected for this study, sign up for an informed consent form, informed about the details of the procedure and the potential risks before treatment and randomized into 2 treatment groups:

* Group A (F-ESWT group): 3 sessions, one per week, of electromagnetic focused extracorporeal shockwave treatment (3000 impulses at 0.12 mJ/mm2 per session).
* Group B (placebo group): 3 sessions, one per week, of electromagnetic focused extracorporeal shockwave treatment (3000 impulses at 0.01 mJ/mm2 per session).

All treatments will be performed by the senior authors. In all cases, a focused electromagnetic shockwave device will be used (Duolith® SD-1, STORZ Medical, Switzerland).

The procedure will be performed with the patient in lateral positioning of the decubitus pronus. The treatment area will be prepared with a coupling ultrasound gel to minimize the loss of shockwave energy at the interface between the tip of the applicator and the skin. The inline ultrasonic guide will be used to concentrate the shockwaves on the injury area in the muscle. No local anesthesia will be applied.

STUDY EVALUATIONS Injury size: Evaluation of the three major diameters of the lesion. Grade of repair process (A,B,C,D): Evaluation of the repair process with stages from A to D, where A represented the absence of repair, B a start in the repair process with less than 50 % scar tissue, C advanced repair process with more than 50 % repaired tissue and stage D when complete repair was observed.

Visual Analogue Scale (VAS): The visual analogue scale (VAS) is considered to be one of the best methods available for the estimation of the intensity of pain. The VAS provides a continuous scale for magnitude estimation and consists of a straight line, the ends of which are defined in terms of the extreme limits of pain experience. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain experienced. This gives the greatest freedom to choose pain's exact intensity. It also gives the maximum opportunity for each respondent to express a personal response style.

Lower Extremity Functional Scale (LEFS): The Lower Extremity Functional Scale (LEFS) is a sensitive and reliable outcome measure that has commonly been used in patients with hip and knee dysfunction. The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals. The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities.

Tegner activity scale: Tegner activity level scale is a graduated list of activities of daily living, recreation and competitive sports. The patient is asked to select the level of participation that best describes their current level of activity (before injury). The score varies from 0-10. A score of 0 represents sick leave or disability pension, whereas a score of 10 corresponds to participation in national and international elite competitive sports >6 Roles and Maudsley scale: The RM scale is a subjective 4-point patient assessment of pain and limitations of activity. The RM score has been used extensively at centers throughout the world to assess outcome after SWT. On the scale, 1 point indicates an excellent result with the patient having no symptoms. Two points indicate a good result with the patient significantly improved from the pretreatment condition and satisfied with the result. Three points indicate a fair result with the patient somewhat improved from the pretreatment condition and partially satisfied with the treatment outcome. Four points indicate a poor outcome with symptoms identical or worse than the pretreatment condition and dissatisfaction with the treatment result.

Likert scale (1-6): Degree of recovery compared with baseline, measured on a 6-point Likert scale (completely recovered to much worse). Success rates will be calculated by dichotomizing responses.

Return to play: Return to Play is the process of deciding when an injured or ill athlete may safely return to practice or competition.

ETHICS/PROTECTION OF HUMAN SUBJECTS

1. Ethical Standard: This clinical study was designed and shall be conducted and reported in accordance with the International Conference for Harmonization (ICH) Harmonized Tripartite Guidelines for Good Clinical Practice, with applicable local regulations (including European Directive 2001/20/EC), and with the ethical principles laid down in the Declaration of Helsinki.
2. Independent Ethics Committee: The protocol, informed consent form, recruitment materials, and all subject materials will be submitted to an Independent Ethics Committee (IEC) in each center for review and approval. Approval of both the protocol and the consent form must be obtained before any subject is enrolled. The implementation of any change in the protocol will not be permitted until the principal investigator and the IEC have provided written approval of the change.
3. Informed Consent Process: Informed consent is a process that is initiated prior to the individual agreeing to participate in the study and continues throughout study participation. An extensive discussion of the risks and possible benefits of study participation will be held with the subjects. A consent form describing in detail the study procedures and risks will be given to the subject. Consent forms will be IEC-approved, and the subject is required to read and review the document or have the document read to him or her. The investigator or designee will explain the research study to the subject and answer any questions that may arise. The subject will sign the informed consent document prior to any study-related assessments or procedures. Subjects will be given the opportunity to discuss the study with their families and take all the time they need prior to agreeing to participate. They may withdraw consent at any time throughout the course of the study. A copy of the signed informed consent document will be given to the subjects for their records. The rights and welfare of the subjects will be protected by emphasizing to them that the quality of their clinical care will not be adversely affected if they decline to participate in this study. The consent process will be documented in the clinical records.
4. Subject Confidentiality: Subject confidentiality shall be guaranteed at all times by the investigators, study staff, and the sponsor and their delegates. The study protocol, documentation, data, and all other information generated will be strictly confidential. No information concerning the study or the data will be released to any unauthorized third party without prior written approval of the sponsor.

The study monitor or other authorized representatives of the sponsor may inspect all study documents and records required to be maintained by the investigator, including but not limited to the medical records of the study subjects. The clinical study site will permit access to such records.

DATA HANDLING AND RECORD KEEPING The investigator will be responsible for the completeness, accuracy and timeliness of the data reported. All source documents should be completed in a neat, legible manner to ensure the accurate interpretation of data. The Investigator is required to verify the data transcribed onto the database.

The study monitors then have to check the database against the source documents for accuracy and validity as per the monitoring schedule, as applicable.

1. Data Management Responsibilities Data collection and accurate documentation are the responsibility of the study staff under the supervision of the investigator. All source documents and laboratory reports must be reviewed by Site staff and data entry staff, who will ensure that they are accurate and complete. Unanticipated problems and adverse events must be reviewed by the investigator or designee.
2. Protocol Deviations The occurrence of any protocol deviations will be reported during the conduct of the study. All significant protocol deviations will be recorded and reported in the clinical study report.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years old
* Informed consent signed
* Soccer injury
* Diagnosis of acute indirect common tendon of the hamstring injury
* Time of diagnosis < 2 weeks after the injury
* Time to receive the first session of F-ESWT protocol ≤ 2 weeks after the injury

Exclusion Criteria:

* 1 Age < 18 years
* Direct hamstring injury
* Time of diagnosis ≥ 2 weeks after the injury
* Chronic injury or re-injury in the homolateral hamstrings
* Presence of hematoma in the context of the injury
* Injury in a different area than common tendon of the hamstring
* Tumor in the area to be treated
* Wound in the area to be treated
* Anti-inflammatory medication after the injury and/or during the period of treatment
* Coagulation disorders or anticoagulant therapy
* Local infection
* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-29 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Ultrasound evaluation of the injury size | Weekly until recovery (maximum of 10 weeks)
  Evaluation of the three major diameters of the lesion.
Ultrasound evaluation of the injury size | 10 Weekly until recovery (maximum of 10 weeks)
  Evaluation of the repair process with stages from A to D, where A represented the absence of repair, B a start in the repair process with less than 50 % scar tissue, C advanced repair process with more than 50 % repaired tissue and stage D when complete repair was observed.
Return to play period | Weekly until recovery (maximum of 10 weeks)
  Return to Play is the process of deciding when an injured or ill athlete may safely return to practice or competition.

SECONDARY OUTCOMES:
Visual Analogue Scale | Weekly until recovery (maximum of 10 weeks)
  The visual analogue scale (VAS) is considered to be one of the best methods available for the estimation of the intensity of pain. The VAS provides a continuous scale for magnitude estimation and consists of a straight line, the ends of which are defined in terms of the extreme limits of pain experience. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain experienced. This gives the greatest freedom to choose pain's exact intensity. It also gives the maximum opportunity for each respondent to express a personal response style. VAS data of this type is recorded as the number of millimeters from the left of the line with the range 0-100.
Lower Extremity Functional Scale | Weekly until recovery (maximum of 10 weeks)
  The Lower Extremity Functional Scale (LEFS) is a sensitive and reliable outcome measure that has commonly been used in patients with hip and knee dysfunction. The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals. The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention.
Tegner activity scale | Weekly until recovery (maximum of 10 weeks)
  Tegner activity level scale is a graduated list of activities of daily living, recreation and competitive sports. The patient is asked to select the level of participation that best describes their current level of activity (before injury). The score varies from 0-10. A score of 0 represents sick leave or disability pension, whereas a score of 10 corresponds to participation in national and international elite competitive sports >6. Score can only be achieved if the person participates in recreational or competitive sport.
Roles and Maudsley scale | Weekly until recovery (maximum of 10 weeks)
  The RM scale is a subjective 4-point patient assessment of pain and limitations of activity. The RM score has been used extensively at centers throughout the world to assess outcome after SWT. On the scale, 1 point indicates an excellent result with the patient having no symptoms. Two points indicate a good result with the patient significantly improved from the pretreatment condition and satisfied with the result. Three points indicate a fair result with the patient somewhat improved from the pretreatment condition and partially satisfied with the treatment outcome. Four points indicate a poor outcome with symptoms identical or worse than the pretreatment condition and dissatisfaction with the treatment result.
Likert scale | Weekly until recovery (maximum of 10 weeks)
  Degree of recovery compared with baseline, measured on a 6-point Likert scale (completely recovered to much worse). Success rates will be calculated by dichotomizing responses. Subjects who will report themselves completely recovered or much improved will be counted as successes, and subjects who will report themselves somewhat improved, same, worse, or much worse will be counted as failures.

CONTACTS AND LOCATIONS:
Overall Officials: Montse Garcia, Study Chair — Fundación García Cugat
Locations (1):
- Fundacion Garcia Cugat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No